CLINICAL TRIAL: NCT01373164
Title: A Phase 1b/2 Study With Gemcitabine and LY2157299 for Patients With Metastatic Cancer (Phase 1b) and Advanced or Metastatic Unresectable Pancreatic Cancer (Phase 2)
Brief Title: A Study in Metastatic Cancer and Advanced or Metastatic Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13663; H9H-MC-JBAJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2017-01

CONDITIONS: Neoplasms; Neoplasm Metastasis; Pancreatic Cancer
Keywords: Neoplasms; Neoplasm Metastasis; Pancreatic Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Pancreatic Neoplasms | interventions — LY-2157299; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase 1b: 80 mg Galunisertib + Gemcitabine (Experimental): Cohort 1: 40 mg Galunisertib was administered orally twice daily (BID) for 14 days followed by 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks.
  Interventions: Drug: Galunisertib; Drug: Gemcitabine
- Phase 1b: 160 mg Galunisertib + Gemcitabine (Experimental): Cohort 2: 80 mg Galunisertib was administered orally twice daily for 14 days followed by 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks.
  Interventions: Drug: Galunisertib; Drug: Gemcitabine
- Phase 1b: 300 mg Galunisertib + Gemcitabine (Experimental): Cohort 3: 150 mg Galunisertib was administered orally twice daily for 14 days followed by 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks.
  Interventions: Drug: Galunisertib; Drug: Gemcitabine
- Phase 2: Recommended dose of Galunisertib + Gemcitabine (Experimental): Galunisertib recommended dose (300 mg) determined from phase 1, administered orally twice daily for 14 days followed by 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks.
  Interventions: Drug: Galunisertib; Drug: Gemcitabine
- Phase 2: Placebo + Gemcitabine (Experimental): Placebo administered orally twice daily for 14 days followed 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks.
  Interventions: Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Galunisertib — Administered orally
  Other Names: LY2157299
  Arms: Phase 1b: 160 mg Galunisertib + Gemcitabine; Phase 1b: 300 mg Galunisertib + Gemcitabine; Phase 1b: 80 mg Galunisertib + Gemcitabine; Phase 2: Recommended dose of Galunisertib + Gemcitabine
Drug: Gemcitabine — Administered intravenously
  Other Names: Gemzar; LY188011
Drug: Placebo — Administered orally
  Arms: Phase 2: Placebo + Gemcitabine

SUMMARY:
Phase 1b: To determine the safe and tolerable dose of galunisertib in combination with gemcitabine in patients with solid malignancy

Phase 2a: To compare the overall survival (OS) of patients with Stage II to IV unresectable pancreatic cancer when treated with a combination of galunisertib and gemcitabine with that of gemcitabine plus placebo.

ELIGIBILITY:
Inclusion Criteria: For both Phase 1b and Phase 2 (unless specified in the following), patients are eligible to be included in the study only if they meet all of the following criteria:

For Phase 1b:

* Have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic disease; that is refractory to standard therapy and/or therapies known to provide clinical benefit or for which no standard therapy exists; and/or in which gemcitabine therapy at the proposed doses and schedule would be considered appropriate treatment for the metastatic disease (eg, pancreatic cancer)
* Patients may have received prior chemotherapy, radiotherapy, cancer-related hormone therapy, or other investigational therapy as treatment. There is no limit in the number of previous lines of therapy.

For Phase 1b and Phase 2:

* Have measurable disease or non-measurable disease, defined according to Response Evaluation Criteria In Solid Tumors (RECIST)
* Have given written informed consent prior to any study-specific procedures
* Have adequate organ function including: Hematologic: absolute neutrophil count (ANC) greater than or equal to 1.5 x 10^9/L, platelets greater than or equal to 100 x 10^9/L, and hemoglobin greater than or equal to 9 g/dL. Hepatic: bilirubin less than or equal to 1.5 times upper limit of normal (ULN), and alkaline phosphatase (ALP), aspartate aminotransferase (AST), alanine aminotransferase (ALT)less than or equal to 2.5 times ULN. If the liver has tumor involvement, AST less than or equal to 5 times ULN and ALT less than or equal to 5 times ULN are acceptable. Patients may have endoscopic or radiologic stenting to treat biliary obstructions. If so, then bilirubin must return to less than or equal to 1.5 times ULN and ALP, AST, and ALT to less than or equal to 5 times ULN prior to enrollment. Renal: serum creatinine within normal limits, less than or equal to 1.5 times ULN.
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Patients must have recovered from any Grade 3/4 toxicities of previous therapies
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Prior radiation therapy for treatment of cancer is allowed to <25% of the bone marrow, and patients must have recovered from the acute toxic effects of their treatment prior to study enrollment. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study entry.
* Male and female patients with reproductive potential must use an approved contraceptive method during and for 3 months after discontinuation of study treatment. Women of childbearing potential must have a negative beta-human chorionic gonadotropin (B-HCG) pregnancy test documented within 14 days prior to treatment. If condoms are used as a barrier contraceptive, a spermicidal agent should be added to ensure that pregnancy does not occur. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

For Phase 2:

* Have histological or cytological diagnosis of adenocarcinoma of the pancreas that is locally advanced (Stage II, III) or metastatic (Stage IV) and not amenable to resection with curative intent. Patients with previous radical surgery for pancreatic cancer are eligible after progression is documented. If they received adjuvant chemotherapy or chemoradiotherapy with gemcitabine, they can be enrolled if the treatment was completed 3 months before or longer
* Tumor tissue or unstained slides are available from original biopsy or resection or other tumor biopsies
* Patients may have received previous adjuvant treatment with gemcitabine with or without radiotherapy for pancreatic cancer. Adjuvant treatment must have finished at least 6 months before enrolling.

Exclusion Criteria: Patients will be excluded from the study if they meet any of the following criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or unapproved use of a drug or device (other than the investigational product used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have moderate or severe cardiac disease:
* Myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension
* Major abnormalities documented by echocardiography with Doppler (for example, moderate or severe heart valve function defect and/or left ventricular ejection fraction (LVEF) <50%, evaluation based on the institutional lower limit of normal)
* Predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress (for example, family history of aneurysms, Marfan-Syndrome, bicuspid aortic valve, evidence of damage to the large vessels of the heart documented by CT scan or MRI with contrast)
* Are unable to swallow tablets or capsules
* Are pregnant or breastfeeding
* Have any significant medical illnesses that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* Have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ), unless in complete remission and off of all therapy for that disease for a minimum of 3 years
* Have active infection that would interfere with the study objectives or influence study compliance
* Phase 2 only: Endocrine pancreatic tumors or ampullary cancer
* Patients with acute or chronic leukemia or with any other disease likely to have a significant bone marrow infiltration (screening not required)
* Have previously completed or withdrawn from this study or any other study investigating galunisertib or any other TGF-ß inhibitor
* Have known allergy to galunisertib or gemcitabine or any ingredient of galunisertib or gemcitabine formulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-06; Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- United States (3):
  - Florida Hospital Tampa HPG and Foregut Surgery, Tampa, Florida
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liège
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besançon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clermont-Ferrand
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montbéliard
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Friedrichshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mönchengladbach
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reutlingen
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Verona
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

REFERENCES:
- [Derived] Smith CL, Thomas Z, Enas N, Thorn K, Lahn M, Benhadji K, Cleverly A. Leveraging historical data into oncology development programs: Two case studies of phase 2 Bayesian augmented control trial designs. Pharm Stat. 2020 May;19(3):276-290. doi: 10.1002/pst.1990. Epub 2020 Jan 5. PMID 31903699
- [Derived] Melisi D, Garcia-Carbonero R, Macarulla T, Pezet D, Deplanque G, Fuchs M, Trojan J, Kozloff M, Simionato F, Cleverly A, Smith C, Wang S, Man M, Driscoll KE, Estrem ST, Lahn MMF, Benhadji KA, Tabernero J. TGFbeta receptor inhibitor galunisertib is linked to inflammation- and remodeling-related proteins in patients with pancreatic cancer. Cancer Chemother Pharmacol. 2019 May;83(5):975-991. doi: 10.1007/s00280-019-03807-4. Epub 2019 Mar 18. PMID 30887178

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died from any cause and participants who were alive and on study (either on study treatment or in long term follow-up) at study conclusion.
Groups:
- Phase 1b: 80 mg (Milligrams) Galunisertib + Gemcitabine: Cohort 1: 40 mg Galunisertib was administered orally twice daily (BID) for 14 days followed by 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 (milligrams per square meter) was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks.
- Phase 2: 300 mg Galunisertib + Gemcitabine: Galunisertib recommended dose (300 mg) determined from phase 1, administered orally twice daily for 14 days followed by 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks.
Period: Overall Study
Arm/Group | Phase 1b: 80 mg (Milligrams) Galunisertib + Gemcitabine | Phase 1b: 160 mg Galunisertib + Gemcitabine | Phase 1b: 300 mg Galunisertib + Gemcitabine | Phase 2: 300 mg Galunisertib + Gemcitabine | Phase 2: Placebo + Gemcitabine
Started | 5 | 4 | 5 | 104 | 52
Received at Least One Dose | 5 | 4 | 5 | 103 | 52
Completed | 5 | 3 | 4 | 92 | 50
Not Completed | 0 | 1 | 1 | 12 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 10 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Phase 2: Placebo + Gemcitabine: Placebo administered orally twice daily for 14 days followed 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks. participants may continue until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: 80 mg Galunisertib + Gemcitabine | Phase 1b: 160 mg Galunisertib + Gemcitabine | Phase 1b: 300 mg Galunisertib + Gemcitabine | Phase 2: 300 mg Galunisertib + Gemcitabine | Phase 2: Placebo + Gemcitabine | Total
Number analyzed (Participants) | 5 | 4 | 5 | 103 | 52 | 169
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (12.9) | 63.8 (9.0) | 56.6 (9.2) | 67.3 (8.2) | 66.3 (8.9) | 63.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 46 | 24 | 76
  Male | 5 | 1 | 2 | 57 | 28 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 4 | 4 | 37 | 18 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 66 | 34 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 0 | 2
  White | 3 | 4 | 5 | 95 | 50 | 157
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 8 | 2 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 0 | 0 | 0 | 4 | 2 | 6
  United States | 5 | 2 | 1 | 7 | 4 | 19
  Italy | 0 | 0 | 0 | 23 | 10 | 33
  France | 0 | 0 | 0 | 21 | 9 | 30
  Germany | 0 | 0 | 0 | 22 | 14 | 36
  Spain | 0 | 2 | 4 | 26 | 13 | 45

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Recommended Phase 2 Dose
Description: The recommended Phase 2 dose was the highest dose where less than 1/3 of participants experienced dose limiting toxicities (DLTs). The recommended dose was determined based on a review of overall toxicity, dose reductions, omissions, and pharmacokinetic information from Phase 1b.
Time Frame: Time of first phase 1b dose until time of last phase 1b dose (up to 1 year)
Population: Phase 1b: All participants who received at least one dose of study drug.
Measure: Number; unit: milligrams (mg)
Groups:
- Phase 1b Participants: Participants received galunisertib at a starting dose of 80 mg/day in combination with gemcitabine. Dose escalation proceeded in cohorts of between 3 to 6 evaluable participants until ≥2 participants experienced a dose limiting toxicity (DLT) or an galunisertib dose level of 300 mg/day was reached.
Arm/Group | Phase 1b Participants
Number analyzed (Participants) | 14
milligrams (mg) | 300

2. Primary Outcome: Phase 2: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death from any cause. For each participant who is not known to have died as of the data-inclusion cut-off date for a particular analysis, overall survival duration was censored for that analysis at the date of last prior contact.
Time Frame: Baseline to date of death from any cause (up to 2 years)
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline observation. Number of participants censored were Galunisertib + Gemcitabine = 20 and Placebo + Gemcitabine = 4.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 2: Placebo + Gemcitabine: Placebo administered orally twice daily for 14 days followed 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks. Participant's may continue until disease progression, unacceptable toxicity, or another withdrawal criterion is met.
Arm/Group | Phase 2: 300 mg Galunisertib + Gemcitabine | Phase 2: Placebo + Gemcitabine
Number analyzed (Participants) | 104 | 52
Months | 8.9 [7.3 to 11.1] | 7.1 [5.8 to 9.0]
Statistical Analysis 1: Comparison: Phase 2: 300 mg Galunisertib + Gemcitabine vs Phase 2: Placebo + Gemcitabine; Test type: Superiority — The planned primary analysis for this study utilized a Bayesian exponential-likelihood model, incorporating historical overall survival (OS) data from 2 studies (Oettle et al. 2005; Saif et al. 2009). The primary analysis was performed using strong borrowing from the historical data. The model was estimated to borrow approximately 37 events from the historical studies; Bayesian Analysis; Primary comparison was to be considered successful if there was at least 0.85 posterior probability that the hazard ratio (HR) for OS of LY+Gem is <1; Hazard Ratio (HR) = 0.794, 95% CI 2-sided [0.590 to 1.085] — This is a Credible Interval estimated from the Bayesian analysis

3. Secondary Outcome: Phase 1b: Pharmacokinetics: Area Under the Concentration-Time Curve at Steady State From Time Zero to 24 Hours (AUC[0-24], ss) and Time Zero to Infinity (AUC[0-∞], ss)
Description: AUC[0-24h] is a combined measure obtained from Day 14 at 0 hour (pre-dose), 0.5, 2,3, 6 hours post dose and morning doses from 24h and 48h to compute. AUC0-infinity will take 48h and extrapolation beyond this in addition to earlier time points to be calculated. All mentioned time points are used to calculate the two AUCs.
Time Frame: Cycle 1 Days 14 (predose; 0.5, 2, 3, and 6 hours post dose), 24h (Days 15) and 48h (Days 16)
Population: Phase 1b: All participants who received at least one dose of study drug and had evaluable PK (pharmacokinetics) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Phase 1b: 80 mg Galunisertib + Gemcitabine | Phase 1b: 160 mg Galunisertib + Gemcitabine | Phase 1b: 300 mg Galunisertib + Gemcitabine
Number analyzed (Participants) | 3 | 2 | 3
nanogram*hour per milliliter (ng*h/mL)
  AUC(0-24) | 2530 (116) | NA (NA) — Not analyzed due to insufficient number of participants with enough PK samples. | 9090 (27)
  AUC(0-∞) | 2740 (117) | NA (NA) — Not analyzed due to insufficient number of participants with enough PK samples. | 10600 (10)

4. Secondary Outcome: Phase 1b: Pharmacokinetics: Maximum Plasma Drug Concentration at Steady State (Cmax,ss)
Description: Plasma samples for pharmacokinetic (PK) analysis were obtained on Day 14 at 0 hours (Pre-dose), 0.5, 2, 3, 6 hours post dose and morning doses from 24h and 48h. Cmax takes all time points post dose into account and one value is reported.
Time Frame: Cycle 1 Days 14 (predose; 0.5, 2, 3, and 6 hours post dose), 24h (Days 15) and 48h (Days 16)
Population: Phase 1b: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1b: 80 mg Galunisertib + Gemcitabine | Phase 1b: 160 mg Galunisertib + Gemcitabine | Phase 1b: 300 mg Galunisertib + Gemcitabine
Number analyzed (Participants) | 3 | 2 | 3
nanogram per milliliter (ng/mL) | 385 (101) | NA (NA) — Not analyzed due to insufficient number of participants with enough PK samples. | 1050 (39)

5. Secondary Outcome: Phase 1b: Number of Participants With Tumor Response
Description: Response was defined using RECIST (Response Evaluation Criteria in Solid Tumors) version 1.1. Complete Response (CR) was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; Partial Response (PR) was defined as having at least a 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD) was defined as having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir; Stable Disease (SD) was defined as small changes that did not meet above criteria.
Time Frame: Baseline to end of Phase 1b (up to 1 year)
Population: Phase 1b: All participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Phase 1b: 80 mg Galunisertib + Gemcitabine | Phase 1b: 160 mg Galunisertib + Gemcitabine | Phase 1b: 300 mg Galunisertib + Gemcitabine
Number analyzed (Participants) | 5 | 4 | 5
Participants
  Progressive Disease (PD) | 3 | 1 | 2
  Stable Disease (SD) | 1 | 2 | 2
  Partial Response (PR) | 0 | 1 | 0
  Non-Complete Response/Non-Progressive Disease (NC) | 0 | 0 | 1
  Not Assessed (NA) | 1 | 0 | 0

6. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS is defined as the date of randomization to the first date of progression of disease or of death from any cause. For each participant who is not known to have died or to have had a progression of disease as of the data-inclusion cut-off date for a particular analysis, PFS will be censored at the date of last prior contact. PFS will be calculated and analyzed twice: (1) including clinical progressions of disease not based on lesion measurements, and (2) excluding clinical progressions. Progression Disease (PD) was defined as having at least a 25% increase in the sum of the longest diameter of target lesions.
Time Frame: Baseline to first date of progressive disease or death due to any cause (up to 2 years)
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline observation. Number of participants censored were Galunisertib + Gemcitabine = 21 and Placebo + Gemcitabine = 11.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: 300 mg Galunisertib + Gemcitabine | Phase 2: Placebo + Gemcitabine
Number analyzed (Participants) | 104 | 52
Months | 4.11 [2.66 to 5.42] | 2.86 [1.94 to 3.75]

7. Secondary Outcome: Phase 2: Percentage Change From Baseline in Tumor Size (CTS)
Description: Change in tumor size is defined as the maximum percent change from baseline in the sum of target lesions. Change was assessed in each participant using radiographic imaging.
Time Frame: Baseline, end of Cycle 2 (up to 56 days)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for change in tumor size.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change in tumor size
Arm/Group | Phase 2: 300 mg Galunisertib + Gemcitabine | Phase 2: Placebo + Gemcitabine
Number analyzed (Participants) | 104 | 52
Percent change in tumor size
  Independent Assessor 1: number analyzed (Participants) | 70 | 35
  Independent Assessor 1 | 0.95 [0.90 to 1.01] | 0.92 [0.87 to 0.98]
  Independent Assessor 2: number analyzed (Participants) | 66 | 33
  Independent Assessor 2 | 1.03 [0.95 to 1.11] | 0.98 [0.92 to 1.05]

8. Secondary Outcome: Phase 2: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate[ORR])
Description: Overall response rate is the best response of complete response (CR) or partial response (PR) as classified by the independent central review according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline to measured progressive disease (up to 2 years)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for ORR.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: 300 mg Galunisertib + Gemcitabine | Phase 2: Placebo + Gemcitabine
Number analyzed (Participants) | 104 | 52
Percentage of Participants | 10.6 [5.4 to 18.1] | 3.8 [0.5 to 13.2]

9. Secondary Outcome: Phase 2: Population Pharmacokinetics (PK): Area Under the Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24])
Description: AUC[0-24] is a combined measure obtained from Day 14 at 0 hour (pre-dose), 0.5, 2,3, 6 hours post dose and morning doses from 24h and 48h to compute.
Time Frame: Cycle 1 Days 14 (predose; 0.5, 2, 3, and 6 hours post dose), 24h (Days 15) and 48h (Days 16)
Population: All randomized participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Mean (Inter-Quartile Range); unit: mg*h/L
Arm/Group | Phase 2: 300 mg Galunisertib + Gemcitabine
Number analyzed (Participants) | 99
mg*h/L | 5.56 [3.82 to 7.91]

10. Secondary Outcome: Phase 2: Population PK: Maximum Concentration (Cmax) of Galunisertib
Description: as for outcome 4
Time Frame: Cycle 1 Days 14 (predose; 0.5, 2, 3, and 6 hours post dose), 24h (Days 15) and 48h (Days 16)
Population: All randomized participants who received at least 1 dose of study drug with evaluable PK data.
Measure: Mean (Inter-Quartile Range); unit: ng/mL
Arm/Group | Phase 2: 300 mg Galunisertib + Gemcitabine
Number analyzed (Participants) | 99
ng/mL | 904 [668 to 1194]

11. Secondary Outcome: Phase 2: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) at Study Completion
Description: The BPI-SF Pain Severity Subscale was a participant-rated questionnaire that measured the severity of pain. Severity scores could have ranged from 0 (no pain) to 10 (pain as bad as you can imagine) for questions that included assessing average pain in the past 24 hours.
Time Frame: Baseline, study treatment completion (up to 1 year)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for BPI-sf.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo+Gemcitabine: Placebo administered orally twice daily for 14 days followed 14 days of rest (28 day cycle).
  Gemcitabine at a dose of 1000 mg/m^2 was administered intravenously once per week for 7 weeks followed by 1 week of rest and then once per week for 3 weeks of every 4 weeks.
Arm/Group | Phase 2: 300 mg Galunisertib + Gemcitabine | Placebo+Gemcitabine
Number analyzed (Participants) | 7 | 2
Units on a scale | 2.54 (2.53) | 1.50 (2.12)

12. Secondary Outcome: Phase 2: Change From Baseline in Carbohydrate Antigen 19.9 (CA19-9) Level at First Study Completion Follow-up
Description: Carbohydrate antigen 19-9 (CA 19-9) is a modified Lewis(a) blood group antigen, and has been used as a tumor marker. The outcome measure is the median, minimum and maximum values from participants who had samples collected at baseline and at follow-up
Time Frame: Baseline, study treatment completion after first follow up visit (up to 1 year)
Population: All randomized participants who received at least 1 dose of study drug and had baseline and a post-baseline measurement for CA19-9 level.
Measure: Median (Full Range); unit: Units/Milliliter (U/mL)
Arm/Group | Phase 2: 300 mg Galunisertib + Gemcitabine | Phase 2: Placebo + Gemcitabine
Number analyzed (Participants) | 38 | 21
Units/Milliliter (U/mL) | 32.7 [-93.8 to 3636.3] | -33.3 [-98.1 to 2460.9]

ADVERSE EVENTS:
Time Frame: Up to 30 days
Description: All participants who received at least one dose of study drug.
Arm/Group | Phase 1b: 80 mg Galunisertib + Gemcitabine | Phase 1b: 160 mg Galunisertib + Gemcitabine | Phase 1b: 300 mg Galunisertib + Gemcitabine | Phase 2: 300 mg Galunisertib + Gemcitabine | Phase 2: Placebo + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 2/5 | 56/103 | 26/52
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 5/5 | 100/103 | 49/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: 80 mg Galunisertib + Gemcitabine (N=5) | Phase 1b: 160 mg Galunisertib + Gemcitabine (N=4) | Phase 1b: 300 mg Galunisertib + Gemcitabine (N=5) | Phase 2: 300 mg Galunisertib + Gemcitabine (N=103) | Phase 2: Placebo + Gemcitabine (N=52)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 3 (4)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 2 (2)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic pseudocyst drainage (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: 80 mg Galunisertib + Gemcitabine (N=5) | Phase 1b: 160 mg Galunisertib + Gemcitabine (N=4) | Phase 1b: 300 mg Galunisertib + Gemcitabine (N=5) | Phase 2: 300 mg Galunisertib + Gemcitabine (N=103) | Phase 2: Placebo + Gemcitabine (N=52)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 3 (4) | 44 (95) | 28 (35)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (8)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 3 (3) | 34 (76) | 17 (42)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (5) | 1 (1) | 29 (83) | 13 (21)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 26 (38) | 12 (16)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 12 (16) | 5 (6)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (8) | 0 (0) | 13 (14) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1) | 30 (31) | 15 (22)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 23 (56) | 12 (26)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 3 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 4 (9) | 39 (69) | 17 (30)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (4) | 3 (4) | 27 (57) | 19 (26)
Asthenia (General disorders) | 0 (0) | 1 (1) | 3 (4) | 36 (72) | 17 (30)
Chills (General disorders) | 1 (4) | 0 (0) | 0 (0) | 10 (12) | 4 (6)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (4) | 1 (1) | 21 (28) | 9 (14)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 4 (4)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 1 (1) | 23 (33) | 12 (15)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (3) | 3 (8) | 2 (4) | 38 (93) | 11 (17)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 3 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 10 (14) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 8 (14) | 2 (4)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 8 (8) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 11 (31) | 5 (10)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 17 (38) | 8 (14)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 9 (16) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 30 (42) | 13 (18)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (14) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 13 (17) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 0 (0) | 5 (6) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (9) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 6 (7) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (7) | 4 (7)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 6 (6) | 6 (8)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (6) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (10) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (7) | 5 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days